CLINICAL TRIAL: NCT01046929
Title: Clinical Study of Limonene in Women With a Recent Diagnosis of Early Stage Breast Cancer Electing to Undergo Excision Surgery
Brief Title: Limonene Study in Women With Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sherry Chow, Research Professor of Medicine, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UAz 09-0447-04; 1R21CA123033-01A2 (NIH)
Record Dates: First submitted 2010-01-08; First posted 2010-01-12 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: limonene; breast cancer; cancer prevention
MeSH Terms: conditions — Breast Neoplasms | interventions — Limonene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- limonene (Experimental)
  Interventions: Dietary Supplement: limonene

INTERVENTIONS:
Dietary Supplement: limonene — oral dosing at 2 gram QD

SUMMARY:
Limonene is a major component in the essential oils of citrus fruits. It has demonstrated promising breast cancer preventive and therapeutic effects in preclinical model systems. This early phase clinical study will evaluate the distribution of limonene to the breast tissue and its associated biological activities after 2 to 6 weeks of limonene dosing in women with a recent diagnosis of early stage breast cancer. This study will help evaluate the potentials of developing limonene as a breast cancer preventive agent.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18 years of age or older
* Women electing to undergo excision surgery for early stage breast cancer
* A minimum of 2 weeks from enrollment to definitive surgery
* Underwent core needle biopsy for breast cancer diagnosis
* No clinical evidence of metastatic breast cancer
* ECOG performance status 0-1
* Participants must have normal organ and marrow function
* Women of child-bearing potential must agree to use adequate contraception
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Concurrent chemotherapy or radiation therapy
* Use of selective estrogen receptor modifiers or aromatase inhibitors within the past 3 months or concurrently
* History of other malignancies within the past 5 years excluding non-melanoma skin cancer and cancers confined to organs with removal as only treatment
* Participated in another clinical intervention trial within the past 3 months
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breast-feeding women
* Use of dietary supplement that contains large amounts of d-limonene (such as Heartburn Free with ROH10 and CoQ with d-limonene) within the past 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
breast tissue limonene level | 2 - 6 weeks

SECONDARY OUTCOMES:
drug effect biomarkers in the breast tissue and serum | 2 - 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States